CLINICAL TRIAL: NCT05330676
Title: The MicroRESUS Study: An Observational Study to Examine the Effects of Circulatory Shock and Resuscitation on Microcirculatory Function and Mitochondrial Respiration After Cardiovascular Surgery.
Brief Title: Evaluation of Microcirculatory Function and Mitochondrial Respiration After Cardiovascular Surgery
Acronym: MicroRESUS
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, John Greenwood, Assistant Professor of Emergency Medicine, Anesthesiology & Critical Care, University of Pennsylvania
Other Study IDs: 843614; KL2TR001879 (NIH)
Record Dates: First submitted 2022-04-09; First posted 2022-04-15 (Actual); Results first posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Shock; Cardiovascular Diseases; Critical Illness
Keywords: microcirculation; mitochondrial respiration; circulatory shock; cardiovascular surgery; resuscitation
MeSH Terms: conditions — Shock; Cardiovascular Diseases; Critical Illness | interventions — Coronary Artery Bypass; Replantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood mononuclear cells, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No shock: Patients who have no evidence of clinical malperfusion or require vasoactive agents after cardiac surgery.
  Interventions: Procedure: coronary artery bypass grafting, valve repair/replacement
- Shock: Patients who have evidence of clinical malperfusion or require vasoactive agents after cardiac surgery.
  Interventions: Procedure: coronary artery bypass grafting, valve repair/replacement

INTERVENTIONS:
Procedure: coronary artery bypass grafting, valve repair/replacement — cardiovascular surgery with cardiopulmonary bypass

SUMMARY:
This study will examine the differences in microcirculatory function and mitochondrial respiration in patients with shock after cardiovascular surgery.

DETAILED DESCRIPTION:
Post-cardiotomy shock (PCS) occurs in up to 5% of cardiovascular surgeries and has an in-hospital mortality rate as high as 75%. It is unclear if patients with PCS despite achieving standard resuscitation goals have impairments in oxygen delivery or oxygen utilization. This study will examine the difference in microcirculatory function and mitochondrial respiration in patients with shock to better understand the driving mechanism of bioenergetic failure in patients with PCS.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old)
* Receiving elective coronary artery bypass graft (CABG)
* Receiving valvular surgery requiring cardiopulmonary bypass

Exclusion Criteria:

* Unable to tolerate sublingual microcirculatory flow imaging (e.g., non-intubated patients dependent upon oxygen by facemask, poor mouth opening)
* receiving an emergent procedure
* have an actively treated malignancy
* mitochondrial disorder
* receiving surgery requiring deep hypothermic circulatory arrest.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cardiovascular disease
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C. Greenwood, Principal Investigator — Perelman School of Medicine at the University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The protocol for this trial will be published in a peer reviewed journal. The anonymized dataset supporting the results of this report will be available via the Zenodo research data repository.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Derived] Greenwood JC, Talebi FM, Jang DH, Spelde AE, Gordon EK, Horak J, Acker MA, Kilbaugh TJ, Shofer FS, Augoustides JGT, Brenner JS, Muzykantov VR, Bakker J, Abella BS. Anaerobic Lactate Production Is Associated With Decreased Microcirculatory Blood Flow and Decreased Mitochondrial Respiration Following Cardiovascular Surgery With Cardiopulmonary Bypass. Crit Care Med. 2024 Aug 1;52(8):1239-1250. doi: 10.1097/CCM.0000000000006289. Epub 2024 Apr 5. PMID 38578158

RESULTS

PARTICIPANT FLOW:
Groups:
- Prolonged Organ Dysfunction: Patients with 28 days or less of vasoactive and ventilator free days (VVFDs) at postoperative day 30
  coronary artery bypass grafting, valve repair or replacement; cardiovascular surgery with cardiopulmonary bypass
- No Prolonged Organ Dysfunction: Patients with greater than 28 vasoactive and ventilator free days (VVFDs) at postoperative day 30.
  coronary artery bypass grafting, valve repair/replacement: cardiovascular surgery with cardiopulmonary bypass
Period: Overall Study
Arm/Group | Prolonged Organ Dysfunction | No Prolonged Organ Dysfunction
Started | 38 | 104
Completed | 36 | 95
Not Completed | 2 | 9
Not completed — Inadequate imaging quality for final analysis | 2 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prolonged Organ Dysfunction | No Prolonged Organ Dysfunction | Total
Number analyzed (Participants) | 36 | 95 | 131
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 37 | 52
  >=65 years | 21 | 58 | 79
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 31 | 42
  Male | 25 | 64 | 89
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 30 | 87 | 117
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Perfused Vessel Denisty (PVD)
Description: Perfused vessel density (PVD) was measured with incident darkfield microscopy (units mm/mm^2)
Time Frame: PVD was measured at baseline (immediately prior to surgery), at ICU admission, approximately 4 hours after surgery, then at 24 hours.
Population: Patient met criteria for the primary outcome if they had 28 vasoactive and ventilator free days (VVFDs) or more at postoperative day 30.
Measure: Mean (Standard Deviation); unit: mm/mm^2
Arm/Group | Prolonged Organ Dysfunction | No Prolonged Organ Dysfunction
Number analyzed (Participants) | 36 | 95
mm/mm^2
  Baseline | 22.8 (4.9) | 23.8 (5.2)
  ICU Admission | 20.2 (3.7) | 22.5 (4.7)
  4-hours after surgery | 21.1 (3.9) | 22.8 (4.9)
  24-hours | 22.3 (5.0) | 23.8 (5.2)

ADVERSE EVENTS:
Time Frame: Duration of in-hospital stay, an average of 10 days.
Arm/Group | Prolonged Organ Dysfunction | No Prolonged Organ Dysfunction
All-Cause Mortality (participants affected / at risk) | 3/36 | 5/95
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/95
Other Adverse Events (participants affected / at risk) | 0/36 | 0/95

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT05330676/Prot_SAP_000.pdf